CLINICAL TRIAL: NCT04145076
Title: Can Brain Activation and Connectivity Predict Treatment Response to Two Serotonergic Medications (Citalopram and Tianeptine) in Subjects With Autism Spectrum Disorders (ASD)?
Brief Title: Brain Response to Serotonergic Medications in ASD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Responsible Party: Principal Investigator, Dr Grainne McAlonan, Deputy head of department, King's College London
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 14/LO/0663
Record Dates: First submitted 2019-10-25; First posted 2019-10-30 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Autism Spectrum Disorder
Keywords: citalopram; tianeptine; pharmacological imaging
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Citalopram; tianeptine

STUDY DESIGN:
Intervention Model Description: Repeated-measures cross-over study, where each subject receives each of three pharmacological probes once (order of drug administration was pseudorandomised).
Who Masked: Participant, Investigator
Masking Description: Participants and investigators are blinded to the drug condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Placebo, Citalopram, Tianeptine (Experimental): Dose order: Placebo, Citalopram, Tianeptine
  Interventions: Drug: Placebo; Drug: Citalopram; Drug: Tianeptine
- Placebo, Tianeptine, Citalopram (Experimental): Dose order: Placebo, Tianeptine, Citalopram
  Interventions: Drug: Placebo; Drug: Citalopram; Drug: Tianeptine
- Citalopram, Placebo, Tianeptine (Experimental): Dose order: Citalopram, Placebo, Tianeptine
  Interventions: Drug: Placebo; Drug: Citalopram; Drug: Tianeptine
- Citalopram, Tianeptine, Placebo (Experimental): Dose order: Citalopram, Tianeptine, Placebo
  Interventions: Drug: Placebo; Drug: Citalopram; Drug: Tianeptine
- Tianeptine, Placebo, Citalopram (Experimental): Dose order: Tianeptine, Placebo, Citalopram
  Interventions: Drug: Placebo; Drug: Citalopram; Drug: Tianeptine
- Tianeptine, Citalopram, Placebo (Experimental): Dose order: Tianeptine, Citalopram, Placebo
  Interventions: Drug: Placebo; Drug: Citalopram; Drug: Tianeptine

INTERVENTIONS:
Drug: Placebo — Two oral doses of placebo.
Drug: Citalopram — Single oral dose of citalopram (20mg) and single oral dose of placebo.
Drug: Tianeptine — Single oral dose of tianeptine (12.5mg) and single oral dose of placebo.

SUMMARY:
This study investigates brain response to single acute dose of citalopram, tianeptine, and placebo in males with and without autism spectrum disorder.

DETAILED DESCRIPTION:
There is increasing evidence that the serotonin (5-HT) system is implicated in autism spectrum disorder (ASD), with the standard treatment for depression and anxiety in both the general population and ASD includes targeting the 5-HT system with selective serotonin reuptake inhibitors (SSRIs) citalopram. Some individuals with ASD have a good treatment response but others do not. Tianeptine, which has a different mechanism of action to SSRIs, is also an effective antidepressant. As it is unlikely that all individuals with ASD will respond to the same treatment, the investigators aim to conduct a pharmacological magnetic resonance imaging (phMRI) investigation to elucidate the neural mechanisms underlying the response to citalopram and tianeptine in ASD. The investigators are inviting 50 male adults with ASD and 50 male adults without ASD. Each participant receives each drug once (20 mg citalopram, 12.5 mg tianeptine, or placebo) and MRI is used to obtain measures of brain biochemistry, activity, and connectivity. The investigators also acquire data from questionnaires, electroencephalography, neurocognitive tests and blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Intelligence Quotient (IQ) above 70
* Has capacity and is capable of giving written informed consent
* Able to read, comprehend and record information written in English
* Bodyweight of <120 kg and BMI within the range 18.5 - 33 kg/m2 (inclusive).
* Not taking medication directly affecting gamma-aminobutyric acid (GABA) neurotransmission for at least the past 4 weeks
* Not taking medication directly affecting the serotonergic system for at least the past 4 weeks
* ASD only: Diagnosis of Autism Spectrum Disorder (ICD 10-R criteria, confirmed using the Autism Diagnostic Interview (ADI) and/or ADOS) including atypical autism
* ASD only: Being recommended drug therapy for symptoms of depression and/or anxiety
* Controls only: No diagnosis of Autism Spectrum Disorder (ICD 10-R criteria, confirmed using the ADI and/or ADOS)
* Controls only: No diagnosis of major depressive disorder according to the Diagnostic and Statistical Manual of Mental Disorders (DSM) IV or ICD 10.

Exclusion Criteria:

* Current risk of self-harm
* Acute risk of suicidality (e.g., current suicidal ideations)
* Age < 18 years or > 60 years old.
* Taking medication directly affecting the serotonergic system (e.g. SSRIs, Tricyclic antidepressants)
* Taking medication directly affecting GABA neurotransmission (e.g. antiepileptic drugs, and benzodiazepines)
* Taking antipsychotic medication or medication for attention deficit hyperactivity disorder (ADHD) for the past 4 weeks
* History of dependence to alcohol or substances of abuse (excluding nicotine)
* Major mental illness (e.g. psychosis), or a learning disability (mental retardation)
* Needle phobia
* Medical/genetic disorder associated with ASD
* Diagnosed and treated for hyperkinesis or Tourette's syndrome
* Allergy to food colouring

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-12-15 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Brain excitation and inhibition response to pharmacological stimulation as assessed by magnetic resonance spectroscopy | In the months 1-2 following the last day of scanning
  The measure of brain excitation and inhibition response to placebo, citalopram, and tianeptine includes the following:
  Assessment of the ratio of brain excitation and inhibition (measured as the balance of excitatory and inhibitory neurotransmitters) using proton magnetic resonance spectroscopy.
Brain activation response to pharmacological stimulation as assessed by functional magnetic resonance imaging | In the months 3-4 following the last day of scanning
  The measure of brain activation response to placebo, citalopram, and tianeptine includes the following:
  Assessment of the blood-oxygen-level-dependent activation during tasks using functional magnetic resonance imaging.
Brain connectivity response to pharmacological stimulation as assessed by resting-state functional magnetic resonance imaging | In the months 5-6 following the last day of scanning
  The measure of brain connectivity response to placebo, citalopram, and tianeptine includes the following:
  Assessment of the regional homogeneity during resting-state using functional magnetic resonance imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Grainne McAlonan, PhD, Principal Investigator — King's College London; Declan Murphy, PhD, Study Chair — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No